CLINICAL TRIAL: NCT00002932
Title: Phase II Multi-Institutional Trial of Targeted Supradose Cisplatin Chemoradiation for Stage IV Squamous Cell Carcinoma of the Head and Neck
Brief Title: Cisplatin and Radiation Therapy in Treating Patients With Stage IV Cancer of the Head and Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: RTOG-9615; CDR0000065366
Record Dates: First submitted 1999-11-01; First posted 2004-09-03 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Head and Neck Cancer
Keywords: stage IV squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: cisplatin
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining radiation therapy with chemotherapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of cisplatin and radiation therapy in treating patients with stage IV cancer of the head and neck.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the percentage of patients for whom a complete course of therapy can be administered using targeted supradose cisplatin chemoradiation in patients with squamous cell carcinoma of the head and neck. II. Determine the partial and complete response rate of cisplatin chemoradiation. III. Determine the incidence of adverse events using cisplatin chemoradiation therapy. IV. Determine the rate of disease-free survival and overall survival in these patients. V. Determine the incidence and pattern of recurrence in these patients. VI. Document quality of life measured by disease-specific instruments in these patients.

OUTLINE: All patients receive four courses of cisplatin on days 1, 8, 15, and 22 concurrent with radiotherapy. One course of chemotherapy consists of intra-arterial cisplatin given over 3-5 minutes. Radiotherapy is given 5 days a week for 7 weeks. This weekly cisplatin chemoradiation course will be repeated 4 times, providing recovery from toxicity is present. Dexamethasone is started the evening prior to cisplatin treatment, and continues until the morning following the procedure.

PROJECTED ACCRUAL: 60 patients will be enrolled.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx, or larynx No distant metastatic disease No previous or concurrent head and neck primaries No lip, nasopharynx, or salivary gland lesions No recurrent tumors Stage IV disease comprised of T4 NO-3 lesions

PATIENT CHARACTERISTICS: Age: 18 and over Performance Status: Karnofsky greater than 60 Life Expectancy: Not specified Hematopoietic: ANC greater than 2,000 Platelet count greater than 100,000 Hepatic: Not specified Renal: Creatinine clearance greater than 50 mL/min Cardiovascular: Not specified Other: Not pregnant or nursing No adverse medical illnesses No imaging studies performed greater than one month preregistration No laboratory studies greater than 2 weeks preregistration No other malignancies, except for basal or squamous cell of the skin, within the past 5 years

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy to the head and neck Surgery: No prior surgery to study site other than a biopsy Other: Protocol treatment must begin within 8 weeks of biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 1997-05; Primary Completion 2001-03 (Actual); Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: K. Thomas Robbins, MD, Study Chair — University of Florida
Locations (13):
- United States (13):
  - University of California San Diego Cancer Center, La Jolla, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - CCOP - Baptist Cancer Institute, Memphis, Tennessee
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Vanderbilt Cancer Center, Nashville, Tennessee
  - Fletcher-Allen Health Care, Burlington, Vermont
  - Green Mountain Oncology Group, Rutland, Vermont
  - Naval Medical Center, Portsmouth, Portsmouth, Virginia
  - University Cancer Center, Seattle, Washington
  - University of Washington Neutron Facility and Cancer Center, Seattle, Washington

REFERENCES:
- [Background] Kumar P, Harris J, Garden AS, et al.: Outcome comparisons of four Radiation Therapy Oncology Group (RTOG) trials in patients with stage IV-T4 head and neck (H/N) cancer: encouraging results using intra-arterial (IA) cisplatin (P) and concurrent radiation therapy (RT). [Abstract] J Clin Oncol 22 (Suppl 14): A-5527, 494s, 2004.
- [Result] Robbins KT, Kumar P, Harris J, McCulloch T, Cmelak A, Sofferman R, Levine P, Weisman R, Wilson W, Weymuller E, Fu K. Supradose intra-arterial cisplatin and concurrent radiation therapy for the treatment of stage IV head and neck squamous cell carcinoma is feasible and efficacious in a multi-institutional setting: results of Radiation Therapy Oncology Group Trial 9615. J Clin Oncol. 2005 Mar 1;23(7):1447-54. doi: 10.1200/JCO.2005.03.168. PMID 15735120
- [Result] Targeted chemoradiation (RTOG 96-15) (RADPLAT) for T4 carcinoma of the upper aerodigestive tract: interim analysis of a multi-institutional trial. [Abstract] Proceedings of the International Conference on Head and Neck Cancer A046, 78, 2000.
- [Result] Kumar P, Harris J, Robbins KT, et al.: The feasibility of using intra-arterial cisplatin & radiation therapy for stage IV-T4 head/neck squamous cell carcinoma in a multi-institutional setting: preliminary results of Radiation Therapy Oncology Group (RTOG) trial 9615. Int J Radiat Oncol Biol Phys 48(3 suppl): A-81, 152, 2000.